CLINICAL TRIAL: NCT03636126
Title: Virtual Reality and tACS for Performance Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 018-181
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Law Enforcement Officers

STUDY DESIGN:
Intervention Model Description: The total study time will be 4 weeks. Participants will be asked to use the VR and tACS for two of these four weeks. Participants will be randomly assigned to one of two groups: A) a group that uses the tACS+VR for weeks 1 & 2 or B) a group that uses the tACS+VR for weeks 3 & 4.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- VR + TACS (Experimental): 1. Complete one chapter of the virtual reality game "Land's End" while simultaneously using the tACS system (chapters range in length from approximately 5-20 minutes) after waking up each day (or prior to beginning a work shift).
  2. Use the tACS system without the VR for 20 minutes just before sleep (or at the end of a work shift, whichever time point is most convenient). Table 1. Timeline of Study Treatment
  Interventions: Device: VR + TACS
- No Intervention for 2 Weeks (No Intervention): For 2 weeks of the 4 week study, each group (Group A and Group B) will continue work shifts as usual with no intervention.

INTERVENTIONS:
Device: VR + TACS — TACS- A regulated class of transcranial alternating current stimulation (tACS), called Cranial Electrotherapy Stimulation (CES) by Fisher Wallace Laboratories (FWL) is FDA-Cleared to treat depression, anxiety, and insomnia (Proof of FDA clearance and 510k provided in the appendix). FWL tACS delivers weak non-invasive electrical stimulation (1-4 milliamps at 15, 500, and 15,000 Hz) to the frontal/temporal brain regions by electrodes placed above the temples. Land's End Virtual Reality Game Meta-analyses show Virtual Reality (VR) is an effective non-pharmacological method that reduces obstacles to human performance such as pain, insomnia, anxiety, sleep deprivation, and a variety of other stress responses.
  Arms: VR + TACS

SUMMARY:
The chronic stress of police work may reduce human performance through increases in anxiety, depression, pain, and insomnia. Land's End VR may teach mindful meditation that is associated with reduced anxiety, depression, pain, and insomnia. tACS may produce similar effects to Selective Serotonin Reuptake Inhibitors (SSRIs) without the side effect risks of SSRIs by stimulating neurotransmitter production and modulating the default mode network, resulting in reduced anxiety, depression, pain, and insomnia. These two technologies have not been investigated as interventions among police officers. Therefore, we propose a pilot randomized waitlist-controlled crossover trial of the feasibility and efficacy of Land's End VR and tACS among police officers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* English-Speaking (The measures have not been validated in other languages).
* Willing and able to provide informed consent and participate in the study visit and study follow-up questionnaires
* Able to position head completely upright (90 degrees from the ground) in order to view the entirety of the Virtual Reality video

Exclusion Criteria:

* Hearing or visually impaired where they cannot use the Samsung Gear VR
* History of motion sickness or cyber sickness and unwilling to watch a 10-minute virtual reality video because of it
* Unable to position head completely upright (90 degrees from the ground)
* History of seizures
* Lesions, rashes, or open wounds on face, head, neck, or ears
* Medical device implanted in the head or neck
* Participants with pacemakers
* Participants with known or suspected heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Change in score Assessed at Baseline, 2 weeks and 4 weeks.
  The Numerical Rating Scale (NRS) has been validated as a measure of pain intensity and is one of the most commonly used measures in assessing pain. The NRS asks patients to rate their pain severity on a 0 to 10 scale, with 0 being "no pain" to 10 being "so severe that you can't stand it."
Insomnia Severity Index (ISI) | Change in score Assessed at Baseline, 2 weeks and 4 weeks.
  The Insomnia Severity Index (ISI) is a 7-item, self-report instrument that assesses the severity of insomnia. The ISI has adequate reliability and validity and is frequently used in randomized controlled trials of sleep interventions. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
The Patient Health Questionnaire 8 (PHQ-8) | Change in score Assessed at Baseline, 2 weeks and 4 weeks.
  The PHQ-8 is a brief self-report measure of major depressive disorder. The PHQ-8 is considered to be valid measure of depression for population-based studies and clinical populations with a cut off score of equal or greater than 10 as the diagnostic for current depression. The PHQ-8 is derived from the PHQ-9 by removing the last question regarding suicide assessment.
Primary Care Posttraumatic Stress Disorder Screen (PC-PTSD) | Change in score Assessed at Baseline, 2 weeks and 4 weeks.
  The PC-PTSD is a 4-item"yes" or "no" screen designed for use in medical settings and is the current screening instrument used in the VA system to screen for PTSD. This is considered a psychometrically sound screen for determining the presence and absence of PTSD in the VA setting and has also been used in the civilian primary care population. With a cut-off score of 3, the PC-PTSD has shown 85% diagnostic efficiency, 78% sensitivity, and 87% specificity.
Generalized Anxiety Disorder (GAD7) | Change in score Assessed at Baseline, 2 weeks and 4 weeks.
  The GAD7 is a 7-item questionnaire that measures severity of anxiety. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Therefore, GAD-7 scores range from 0 to 21, with scores of 5, 10, and 15 representing mild, moderate, and severe anxiety symptom levels, respectively

SECONDARY OUTCOMES:
Demographics Questionnaire | Assessed at Baseline
  Participants will be asked to provide standard demographic information (i.e., age, gender, race/ethnicity, level of education, etc.). Participants will also be asked about hearing and visual impairment as well as any history of motion sickness.
Alcohol Use Disorder Identification Test-Consumption (AUDIT-C) | Assessed at Baseline, 2 weeks and 4 weeks.
  Alcohol Use Disorder Identification Test-Consumption (AUDIT-C) is a 3-item alcohol screen that can identify problem alcohol use. The AUDIT-C is scored o a scale of 0-12, each question has 5 answer choices with "a" being 0 points and "e" being 4 points.
Attitudes Toward the Experience Survey | Assessed at 4 weeks
  The Attitudes Toward the Experience Survey is an 8-item NRS that will be used to measure the participant's attitude toward the VR experience. Participants rate the degree to which they agree with the statements on a 1-10 scale, with 0 being "strongly disagree" and 10 being "strongly agree."

CONTACTS AND LOCATIONS:
Locations (1):
- Garland PD, Garland, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided